CLINICAL TRIAL: NCT02441179
Title: Acute Intermittent Hypoxia and Body Weight Supported Treadmill Training: a Potential Therapy for Incomplete Spinal Cord Injury Patients
Brief Title: Acute Intermittent Hypoxia and Body Weight Supported Treadmill Training for Incomplete Spinal Cord Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Pro Ayuda del Niño Lisiado (Other)
Collaborators: Hospital Clinico Mutual de Seguridad (Other)
Responsible Party: Principal Investigator, Angela A Navarrete-Opazo, MD, PhD, Angela A Navarrete-Opazo MD, PhD, Sociedad Pro Ayuda del Niño Lisiado
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0027
Record Dates: First submitted 2015-05-05; First posted 2015-05-12 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-01

CONDITIONS: Spinal Cord Injuries
Keywords: acute intermittent hypoxia; rehabilitation; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acute Intermittent Hypoxia Arm (Experimental): AIH protocol: it consists of 15, 90-second hypoxic episodes (FiO2=0.09) interspersed with 15, 90-second normoxic intervals (FiO2=0.21) for a total time of 45 minutes. This protocol will be repeated every day for 5 consecutive days and then 3 times per week for 3 weeks. Total time: 4 weeks. After this AIH protocol, patients will received body weight-assisted treadmill training (BWSTT) for 45 minutes.
  Interventions: Other: Acute Intermittent Hypoxia; Other: Body weight-assisted treadmill training
- Normoxia Arm (Placebo Comparator): Sham protocol: it consists of continuous normoxia (FiO2=0.21) for 45 minutes for 5 consecutive days and then 3 times per week for 3 weeks. Total time: 4 weeks.After this AIH protocol, patients will received body weight-assisted treadmill training (BWSTT) for 45 minutes.
  Interventions: Other: Body weight-assisted treadmill training; Other: Sham Protocol

INTERVENTIONS:
Other: Acute Intermittent Hypoxia — Patients will breath 9% oxigen for 1.5 minutes interspersed with 1.5 minutes of 21% oxigen (normoxia), 15 times for a total of 45 minutes.
  Arms: Acute Intermittent Hypoxia Arm
Other: Body weight-assisted treadmill training — Patient´s gait will be trained through a weight-assisted treadmill (BWSTT). All recruited patients will start BWSTT at a speed of 0.6 km/hr. The physical therapist will manually correct posture to assure an adequate gait, increasing the speed of treadmill progressively depending upon the patient progress and tolerance. This training will be done immediately after the protocol of AIH or Sham and it will last 45 minutes.
Other: Sham Protocol — It consists of continuous normoxia (FiO2=0.21) for 45 minutes for 5 consecutive days and then 3 times per week for 3 weeks. Total time: 4 weeks.
  Other Names: Placebo Protocol
  Arms: Normoxia Arm

SUMMARY:
Spinal cord injury (SCI) interrupts descending synaptic pathways from brainstem premotor neurons to spinal motor neurons, thereby paralyzing muscles below the neurological level. In recent years, considerable evidence has demonstrated that acute intermittent hypoxia (AIH) elicits plasticity in the spinal cord and strengthens spare synaptic pathways which is expressed as respiratory and somatic functional recovery in animals and humans suffering from incomplete SCI. The fundamental hypothesis guiding this project is that AIH-induced motor plasticity can be "harnessed" to improve walking capacity in incomplete SCI patients, classified as C and D categories according to International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI). The inclusion criteria include patients > 18 years-old, with traumatic or non-traumatic, non-progressive incomplete SCI, onset > 6 months, neurological level C5-T12, with walking ability with or without assistive devices, without joint contractures, orthopedic injuries, osteoporosis, cutaneous lesions, cardiopulmonary complications and a body weight below 150 Kg. A randomized, triple-blind, placebo-controlled parallel design study will be done including 100% of patients fulfilling the criteria. Participants will receive repetitive acute intermittent hypoxia (rAIH: 15 episodes of 90 second 9% inspired oxygen interspersed with 90-second normoxia) or repetitive continued normoxia (rSham: 21% inspired oxygen) combined with 45 minutes body weight-supported treadmill training on 5 consecutive days and then three times per week for 3 weeks. Primary outcome measurement will be the 10-meter walking test. Secondary outcome measurements include the 6-minute walking test, timed up and go test, body/weight load, modified ashworth scale and visual analog scale. All outcomes will be measured before beginning the protocol (baseline), after five days of AIH/Sham (D5), weekly up to the end of the study (W2-W4), and a post-study follow-up for 2 weeks (F1-F2). Aditionally, cognitive assesment before and after the study will be performed using the "Figura compleja de Rey-Osterrieth" and the "Test de aprendizaje verbal España Complutense (TAVEC)". Repetitive AIH and body weight-supported treadmill training may represent a novel, safe, and noninvasive potential therapy to partially restore walking function in incomplete sub-acute and chronic SCI patients, a population with limited, if any, potential for improved function.

DETAILED DESCRIPTION:
Currently, there is no "cure" for spinal cord injuries (SCI). Although the scientific understanding of central nervous system (CNS) regeneration has advanced greatly in the past twenty years, there are still many unknowns with regard to inducing successful regeneration, especially with chronic SCI. A more realistic approach, based on currently available knowledge, to improve the quality of life for a large proportion of the paralyzed population may be to develop treatments that elicit partial functional recovery based on neuroplastic potential of spared neural pathways. In this scenario, acute intermittent hypoxia (AIH) enhances the inherit capacity for neuroplasticity and strengthens surviving synaptic inputs onto spinal motorneurons, which trigger functional recovery following SCI in rats and humans AIH-induced neuroplasticity has been extensively studied in phrenic motor nuclei (C3-C5) through phrenic nerve recording preparations (Mitchell, 2007). Briefly, moderate AIH (3, 5-min hypoxic episodes; PaO2 35-45 mmHg; 5-min intervals) elicits phrenic long term facilitation (pLTF), a type of memory present in the cervical spinal cord. The mechanism of AIH-induced pLTF is that episodic hypoxia activates raphe serotonergic neurons that project to phrenic motor nuclei. Spinal serotonin release during hypoxic episodes subsequently activates serotonin type 2 (5-HT2) receptors coupled to Gq protein on or near phrenic motor neurons, and initiates intracellular cascades that underlie pLTF . pLTF requires spinal 5-HT2 receptor activation , new synthesis of brain-derived neurotrophic factor (BDNF) and activation of its high-affinity receptor tyrosine kinase (TrkB) followed by ERK MAP kinase signaling. Although downstream signaling events from ERK are less clear, it is speculated that glutamate receptors are phosphorylated, increasing glutamatergic transmission and perhaps insertion within phrenic motor neurons, thereby establishing LTF.

Longer time domains of AIH, for example, daily acute intermittent hypoxia (i.e. dAIH, 10 episodes per day, 7 days) have shown to strengthen synaptic pathways to spinal motorneurons and increase respiratory and locomotor recovery after cervical SCI in unanesthetized rats. This functional improvement is accompanied by increased BDNF and TrkB levels within cervical (C7) motor nuclei innervating the forelimb. Although the detailed mechanisms of the functional recovery in somatic thoracic or lumbar motorneurons have not been verified, it has been proposed that the same serotonin-dependent mechanisms facilitate motor output in respiratory and non-respiratory motor nuclei.

The use of dAIH to improve limb function in humans with incomplete, chronic SCI has shown promising results. A single presentation of AIH (15, 1-minute episodes of 9% O2 alternating with 1-minute of 21% O2) in incomplete, chronic (>1 year) spinal cord injury patients, classified as C or D according to the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI), increases the ability to voluntarily generate plantar flexion 4 h post-hypoxia. In a randomized, double-blind, placebo-controlled, crossover design study, the impact of daily AIH (15 episodes per day, 90 sec 9% O2, 60 sec normoxic interval, 5 consecutive days) combined with walking training was studied in 19 chronic, incomplete SCI patients (ISNCSCI D). Daily AIH alone increased walking speed 18% three days after treatment (10 m walk test); whereas dAIH combined with walking training improved both walking speed and distance (37%) after 5 days and 1 week post-dAIH. Importantly, no changes in cognitive function was observed after dAIH, suggesting that this moderate dose of AIH is safe in humans.

Although dAIH (5 consecutive days of AIH) has demonstrated beneficial effects in incomplete SCI patients, its effect last only up to one week; therefore, is important to design extended protocols maintaining the initial functional effect of dAIH over time. Repetitive AIH (rAIH) consisting of AIH three times per week (3×wAIH) for 10 weeks have demonstrated to increase respiratory function and maintain the increased functional effect elicited by dAIH in unanesthetized rats. Moreover, rAIH increases the expression of key molecules involved in AIH-induced spinal plasticity in unanesthetized rats. Therefore, repetitive AIH may represent a safe and effective strategy to enhance functional recovery after chronic incomplete spinal cord injuries.

The protocol of intermittent hypoxia proposed in this project corresponds to a moderate dose of intermittent hypoxia, which is the equivalent of climbing a mountain at 5000 meters altitude. Abundant literature has demonstrated that moderate AIH (≥ 9% O2, < 15 cycles/day) have several multi-systemic beneficial effects: reduces arterial hypertension, strengthens innate immune responses, reduces inflammation, reduces body weight, increases aerobic capacity, improves glucose tolerance, increases bone mineral density, enhances spatial learning and memory, rescues ischemia-induced memory impairment, reduces symptoms of depression, improves post-ischemic recovery of myocardial contractile function, and increases respiratory capacity in chronic obstructive pulmonary disease. Moreover, moderate repetitive AIH improves respiratory and somatic function after SCI, without adverse consequences such as hypertension, neuronal cell loss and/or reactive gliosis or systemic inflammation. Therefore, the potential beneficial effects of AIH are not only limited to spinal cord injuries but include a wide scope of clinical conditions.

Combinatorial therapies, one of them being an activity-based training, can augment plasticity after incomplete SCI. In rats with incomplete SCI, dAIH combined with ladder walking leads to near complete recovery of ladder walking ability. Moreover, dAIH and overground walking improve walking speed and distance in incomplete SCI patients ISNCSCI D. Research studies in animals and humans have found that retraining after SCI using the intrinsic physiologic properties of the nervous system can facilitate the recovery of function. This potential for retraining is based on activity-dependent plasticity driven by repetitive task-specific sensory input to spinal networks.

The most prominent and well-developed activity-based therapy (physical rehabilitation) to date is locomotor training. The fundamental principles of locomotor training are built on the premise of robustly approximating the sensorimotor experience of walking through repetitive practice including: 1) maximize load bearing by the lower extremities and minimize load bearing by the upper extremities, 2) optimize the sensory cues for walking, 3) optimize the kinematics (i.e., trunk and extremities) for each motor task, and 4) maximize recovery strategies and minimize compensatory mechanisms. The fundamental mechanisms supporting this intervention have been derived largely from studies conducted in spinalised animals. Specifically, treadmill training increases axonal regrowth and collateral sprouting proximal to the lesion site in mice (Goldshmit et al., 2008), phosphorylation of Erk1/2 in the motor cortex as well as the spinal cord injury area (Oh et al., 2009), expression of brain-derived neurotrophic factor (BDNF) in the spinal cord, ameliorates muscle atrophy in moderate contused SCI rats, and alters properties of spinal motor neurons. Body weight-supported treadmill training (BWSTT) is based on optimizing sensory inputs relevant to step training, repeated practice, and possible optimization of neuroplasticity. Uncontrolled studies in acute and chronic SCI patients show within-subject improvements in walking ability using BWSTT. Investigators propose that BWSTT therapy provide a behavioral therapy that independently supports positive outcomes.

AIH combined with body weight-assisted training represents a simple and safe, non-pharmacological method for enhancing neuroplasticity in the spinal cord and thus, improving walking function in patients with incomplete spinal cord injuries. At the cellular level, both BWSTT and AIH increase the expression of BDNF. BDNF has a wide repertoire of neurotrophic and neuroprotective properties in the CNS and the periphery; namely, neuronal protection and survival, neurite expression, axonal and dendritic growth and remodeling, neuronal differentiation and synaptic plasticity such as synaptogenesis in arborizing axon terminals, and synaptic transmission efficacy. Thus, BWSTT may serve as a catalyst in tandem with repetitive AIH that when combined develop an even better response.

Currently, there are no approved therapies for chronic SCI; therefore, the approach represents a promising new strategy to enhance function in patients with sub-acute and chronic SCI, where the potential for further functional gains is limited.

Investigators propose a triple blind (patients, outcome assessors and stadistician) randomized, placebo-controlled study testing the combined effect of intermittent hipoxia and body weight-supported treadmill training in incoplete spinal cord injury patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years-old from "Instituto Teletón Santiago" and "Hospital Clínico Mutual de seguridad".
2. C5 to T12 spinal cord injury, classified as ISNCSCI grades C and D
3. Traumatic and non-traumatic, non-progressive lesions
4. Onset > 6 months
5. Ability to ambulate with or without assistive devices
6. Ability to follow verbal or visual commands
7. Signed informed consent

Exclusion Criteria:

1. Orthopedic injuries that are unstable
2. Osteoporosis with high risk of pathological fracture
3. Cutaneous lesions and/or pressure ulcers
4. Joint contractures
5. Cardiopulmonary diseases
6. Body weight exceeding 150 Kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela A Navarrete-Opazo, MD, PhD, Principal Investigator — Instituto de Rehabilitación Infantil Teletón
Locations (2):
- Chile (2):
  - Instituto de Rehabilitación Infantil Teletón, Santiago, Santiago Metropolitan
  - Hospital Mutual de Seguridad, Santiago, Santiago Metropolitan

REFERENCES:
- [Derived] Navarrete-Opazo A, Alcayaga JJ, Sepulveda O, Varas G. Intermittent Hypoxia and Locomotor Training Enhances Dynamic but Not Standing Balance in Patients With Incomplete Spinal Cord Injury. Arch Phys Med Rehabil. 2017 Mar;98(3):415-424. doi: 10.1016/j.apmr.2016.09.114. Epub 2016 Oct 1. PMID 27702556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 67 eligible subjects from 4 hospitals were contacted for screening on site: "Hospital Mutual de seguridad", "Instituto Teletón", "Clínica los Coihues" and "Hospital del Trabajador".Only 38 accepted the invitation.
  The main reason subjects reported to not participate was a tight working schedule and/or lack of employer's permission.
Pre-assignment Details: Out of 38 eligible subjects, three were excluded due to brain trauma history and unknown cognitive deficits.Thus, 35 subjects were enrolled and randomly assigned to the arms.
Groups:
- Acute Intermittent Hypoxia Arm: IH protocol: it consists of 15, 90-second hypoxic episodes (FiO2=0.09) interspersed with 15, 90-second normoxic intervals (FiO2=0.21) for a total time of 45 minutes. This protocol was repeated every day for 5 consecutive days and then 3 times per week for 3 weeks. After each session of IH, patients received body weight-assisted treadmill training (BWSTT) for 45 minutes.
  BWSTT: Patient´s gait was trained through a weight-assisted treadmill (BWSTT). All recruited patients started BWSTT at a speed of 0.6 km/hr. The physical therapist manually corrected posture to assure an adequate gait, increasing the speed of treadmill progressively depending upon the patient progress and tolerance. This training was done immediately after the protocol of IH.
- Normoxia Arm: Sham protocol: it consisted of continuous normoxia (FiO2=0.21) for 45 minutes for 5 consecutive days and then 3 times per week for 3 weeks. After each session, patients received body weight-assisted treadmill training (BWSTT) for 45 minutes.
  BWSTT: Patient´s gait was trained through a weight-assisted treadmill. All recruited patients started BWSTT at a speed of 0.6 km/hr. The physical therapist manually corrected the patient´s posture to assure an adequate gait, increasing the speed of treadmill progressively depending upon the patient progress and tolerance.
Period: Overall Study
Arm/Group | Acute Intermittent Hypoxia Arm | Normoxia Arm
Started | 18 | 17
Completed | 17 | 16
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intermittent Hypoxia Arm: IH protocol: it consists of 15, 90-second hypoxic episodes (FiO2=0.09) interspersed with 15, 90-second normoxic intervals (FiO2=0.21) for a total time of 45 minutes. This protocol was repeated every day for 5 consecutive days and then 3 times per week for 3 weeks. After each session of IH, patients received body weight-assisted treadmill training (BWSTT) for 45 minutes.
  BWSTT: Patient´s gait was trained through a weight-assisted treadmill (BWSTT). All recruited patients started BWSTT at a speed of 0.6 km/hr. The physical therapist manually corrected posture to assure an adequate gait, increasing the speed of treadmill progressively depending upon the patient progress and tolerance. This training was done immediately after the protocol of IH.
- Total: Total of all reporting groups
Arm/Group | Intermittent Hypoxia Arm | Normoxia Arm | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (17) | 42 (17) | 41 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  Chile | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Gait Speed With 10-Meter Walk Test
Description: The 10-meter walk test measures the time (in seconds) that it takes a patient to walk 10m.
Time Frame: Change from baseline in gait speed five days after daily IH.
Population: Analysis was "per protocol"
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Intermittent Hypoxia Arm | Normoxia Arm
Number analyzed (Participants) | 17 | 16
seconds | -10.24 (3.0) | -1.79 (1.75)
Statistical Analysis 1: Comparison: Intermittent Hypoxia Arm vs Normoxia Arm; Test type: Superiority or Other; p = 0.006, Kruskal-Wallis

2. Secondary Outcome: Gait Endurance With the 6-Minute Walk Test
Description: The 6-Minute Walk Test measures the distance (in meters) a patient is able to walk over 6 minutes.
Time Frame: Change from baseline in gait indurance five days after daily IH.
Population: The analysis was "per protocol"
Measure: Mean (Standard Error); unit: meters
Groups:
- Intermittent Hypoxia Arm: IH protocol: it consisted of 15, 90-second hypoxic episodes (FiO2=0.09) interspersed with 15, 90-second normoxic intervals (FiO2=0.21) for a total time of 45 minutes. This protocol was repeated every day for 5 consecutive days and then 3 times per week for 3 weeks. After each session of IH, patients received body weight-assisted treadmill training (BWSTT) for 45 minutes.
  BWSTT: Patient´s gait was trained through a weight-assisted treadmill (BWSTT). All recruited patients started BWSTT at a speed of 0.6 km/hr. The physical therapist manually corrected posture to assure an adequate gait, increasing the speed of treadmill progressively depending upon the patient progress and tolerance. This training was done immediately after the protocol of IH.
Arm/Group | Intermittent Hypoxia Arm | Normoxia Arm
Number analyzed (Participants) | 17 | 16
meters | 43.06 (10.68) | 6.13 (3.41)
Statistical Analysis 1: Comparison: Intermittent Hypoxia Arm vs Normoxia Arm; Test type: Superiority or Other; p = 0.012, Kruskal-Wallis

3. Secondary Outcome: Gait Speed With the Timed up and go Test
Description: The timed up and go test measures the time (in seconds) it takes the patient to stand-up from a seated position in a chair, walk 3 meters at a comfortable and safe pace, turn, walk back to the chair and sit down.
Time Frame: Change from baseline in gait speed five days after daily IH.
Population: The analysis was "per protocol"
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Intermittent Hypoxia Arm | Normoxia Arm
Number analyzed (Participants) | 17 | 16
seconds | -8.71 (3.72) | -2.44 (2.28)
Statistical Analysis 1: Comparison: Intermittent Hypoxia Arm vs Normoxia Arm; Test type: Superiority or Other; p = 0.16, Kruskal-Wallis

4. Secondary Outcome: Percentage of Subjects With Worsening Muscle Tone on the Ashworth Scale
Description: The Ashworth Scale assess muscle tone. It is a 5-points scale ranging from 0 (no increase in muscle tone) to 4 (limb rigid in flexion or extension).
Time Frame: Muscle tone at week 4.
Population: Analysis "per protocol"
Measure: Number; unit: percentage of subjects
Arm/Group | Intermittent Hypoxia Arm | Normoxia Arm
Number analyzed (Participants) | 17 | 16
percentage of subjects | 24 | 31
Statistical Analysis 1: Comparison: Intermittent Hypoxia Arm vs Normoxia Arm; Test type: Superiority or Other; p = 0.57, Chi-squared

5. Secondary Outcome: Percentage of Subjects With Worsening Pain Perception on the "The Visual Analog Test"
Description: The visual analog test assess general pain intensity. It is a 10-score scale ranging from no pain (score 0) to unbearable pain (score 10).
Time Frame: Pain perception at week 4
Population: Analysis "per protocol"
Measure: Number; unit: percentage of subjects
Arm/Group | Intermittent Hypoxia Arm | Normoxia Arm
Number analyzed (Participants) | 17 | 16
percentage of subjects | 11 | 25
Statistical Analysis 1: Comparison: Intermittent Hypoxia Arm vs Normoxia Arm; Test type: Superiority or Other; p = 0.14, Chi-squared

6. Secondary Outcome: Learning and Memory With the Rey-Osterrieth Complex Figure (ROCF) Test
Description: The ROCF is a neuropsychological instrument used for assessment of episodic visual memory.
  Z score ranges from -2 (worse outcome), -1, 0, 1 and 2 (best outcome). The normal population range is between -1 and 1.
  Z score was calculated with the following formula: Z score = (direct score-average for a particular age range)/standard deviation
Time Frame: Episodic visual memory at week 4.
Population: Analysis "per protocol"
Measure: Median (Inter-Quartile Range); unit: Z scores
Arm/Group | Intermittent Hypoxia Arm | Normoxia Arm
Number analyzed (Participants) | 17 | 16
Z scores | 0.19 [-0.84 to 0.49] | 0.16 [-0.30 to 0.60]
Statistical Analysis 1: Comparison: Intermittent Hypoxia Arm vs Normoxia Arm; Test type: Superiority or Other; p = 0.43, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Learning and Memory With the Complutense Verbal Learning Test (TAVEC)
Description: The TAVEC is the Spanish version of the California Verbal Learning Test and is used for the assessment of episodic verbal memory.
  Z score ranges from -2 (worse outcome), -1, 0, 1 and 2 (best outcome). The normal population range is between -1 and 1.
  Z score was calculated with the following formula: Z score = (direct score-average for a particular age range)/standard deviation
Time Frame: Episodic verbal memory at week 4.
Population: Analysis "per protocol"
Measure: Median (Inter-Quartile Range); unit: Z scores
Arm/Group | Intermittent Hypoxia Arm | Normoxia Arm
Number analyzed (Participants) | 17 | 16
Z scores | 0 [-0.5 to 1.0] | 0 [-1 to 0.75]
Statistical Analysis 1: Comparison: Intermittent Hypoxia Arm vs Normoxia Arm; Test type: Superiority or Other; p = 0.55, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Intermittent Hypoxia Arm | Normoxia Arm
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17

LIMITATIONS AND CAVEATS:
Our study included only 4 female subjects; thus, we could not investigate gender differences in response to IH.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No